CLINICAL TRIAL: NCT03953469
Title: Investigating the Short-term Effects of Passiflora Incarnate and Mobile Audio-guided Meditation on Blood Pressure and Heart Rate in Naturopathic Medical Students
Brief Title: Short-term Effects of Passiflora and Meditation on Blood Pressure and Heart Rate
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Bridgeport (Other)
Responsible Party: Principal Investigator, Kimberly Sanders, Principal Investigator, Assistant Professor of Clinical Sciences, University of Bridgeport
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-02-01
Record Dates: First submitted 2019-05-09; First posted 2019-05-16 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Heart Rate Fast; Blood Pressure
Keywords: passionflower; heart rate; blood pressure
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: There are two arms. One arm involves consuming a placebo. The second arm involves taking the Passionflower. Neither the primary investigator nor the participant will know which treatment they are taking.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (No Intervention): (a) Baseline blood pressure readings and one heart rate reading taken after at least 5 minutes of rest time without talking, eating, or caffeine consumption.
  b) will be given 1/4 tsp of blackstrap molasses placebo. Subjects may not consume caffeine or eat food during this time.
  (c) blood pressure readings and one heart rate will be taken 15 minutes after the baseline reading.
- Group II (Active Comparator): 1. Baseline blood pressure readings and one heart rate reading taken after at least 5 minutes of rest time without talking, eating food, or caffeine consumption.
  2. 15 minutes after examination - will be given 1/8 tsp (900mg) of Passiflora incarnata solid extract by Wise Woman Herbals mixed with 1/8 tsp of blackstrap molasses to mask the taste.
  3. blood pressure readings and one heart rate will be taken 15 minutes after the baseline reading.
  Interventions: Dietary Supplement: Passiflora incarnata

INTERVENTIONS:
Dietary Supplement: Passiflora incarnata — One-time administration of 1/8 tsp solid extract Passiflora incarnata providing 900mg of Passiflora incarnata
  Other Names: Passionflower
  Arms: Group II

SUMMARY:
This study is intended to study the effects of one-time acute dosing of a solid extract of Passiflora incarnata, also known as Passionflower, on blood pressure and heart rate in students. Our hypothesis is that blood pressure levels and heart rates will decrease significantly in response to Passiflora incarnata.

ELIGIBILITY:
Inclusion Criteria: all University of Bridgeport students are invited to participate

Exclusion Criteria:

1. Those taking hypertensive medication
2. Those taking anti-anxiety medication, including MAOI medication
3. Those taking blood-thinning medication
4. Those who are pregnant
5. Those who could be pregnant
6. Those who will have surgery 2 weeks before the research date
7. Those who are scheduled to have surgery 2 weeks after the research date
8. Those who have consumed caffeine, food/tyramine containing foods, stimulant medication, cold medicine, decongestant medicine, antihistamine medicine, cough suppressants, alcoholic beverages, or stimulant energy drinks within 2 hours before the study period.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Change in blood pressure between baseline and 15 minutes | 15 minutes
  Change in blood pressure between baseline and 15 minutes
Change in heart rate between baseline and 15 minutes | 15 minutes
  Change in heart rate between baseline and 15 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Sanders, ND, Principal Investigator — University of Bridgeport

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT03953469/Prot_000.pdf
  • Informed Consent Form (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/69/NCT03953469/ICF_001.pdf